CLINICAL TRIAL: NCT04178642
Title: Hepatocellular Carcinoma Under 3 cm Treated by Percutaneous Tumor Destruction: Multicentric Phase 2 Test Evaluating the Impact of Adjuvant Chemotherapy by Intra-arterial Infusion of Idarubicin-lipiodol on the Hepatic Recurrence
Brief Title: The Impact on Hepatic Recurrence After Adjuvant Chemotherapy With Intraarterial Infusion of Idarubicin-Lipiodol
Acronym: LIDA-ADJ
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: no participants enrolled
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RECHMPL19_0073; 2019-001362-15 (EudraCT Number); 7773 (Other: UH Montpellier)
Record Dates: First submitted 2019-11-04; First posted 2019-11-26 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-08

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Intervention Model Description: Prospective multi-center phase II, randomized, unmasked comparative study (ratio 1:1), evaluating the efficacy of an adjuvant treatment by hepatic arterial chemo-infusion of Idarubicin-Lipiodol (experimental group) after percutaneous tumor ablation of hepatocellular carcinoma of size less than 3 cm, versus the absence of adjuvant treatment (standard group), on hepatic recurrence at 1 year.
  It is planned to include 138 patients with hepatocellular carcinoma (CHC) less than 3 cm, non-metastatic, with cirrhosis graded A / B7 on Child Pugh scoring system, and receiving treatment by percutaneous tumor destruction.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- (experimental group) (Experimental): Evaluating the efficacy of an adjuvant treatment by hepatic arterial chemo-infusion of Idarubicin-Lipiodol (experimental group)
  Interventions: Drug: percutaneous destruction of the tumor + Idarubicin-Lipiodol treatment
- (standard group) (Active Comparator): The absence of adjuvant treatment (standard group).
  Interventions: Procedure: Percutaneous destruction of the tumor

INTERVENTIONS:
Drug: percutaneous destruction of the tumor + Idarubicin-Lipiodol treatment — Patients will receive the standard treatment protocol consisting of a percutaneous destruction of the tumor. In addition they will receive an adjuvant treatment by hepatic arterial chemo-infusion of Idarubicin (Zavedos®, Pfizer), which is an anthracycline antineoplastic agent, mixed with Lipiodol (Lipiodol Ultra-Fluid®, Guerbet), which is a contrast agent.
  Arms: (experimental group)
Procedure: Percutaneous destruction of the tumor — Patients will received the standard treatment protocol consisting of a percutaneous destruction of the tumor.
  Arms: (standard group)

SUMMARY:
The aim of this study is to test whether the realization of 3 courses of intra-arterial chemotherapy of idarubicin-lipiodol without embolization, administered non-selectively in the hepatic artery, following the percutaneous tumour ablation of a hepatocellular carcinoma, could constitute an effective adjuvant treatment to reduce the rates of local and intrahepatic distant recurrence and thus improve the survival without hepatic progression.

DETAILED DESCRIPTION:
During this study percutaneous tumor destruction treatment with adjuvant chemotherapy (infusion of Idarubicin-Lipiodol intra-arterial hepatic) will be tested. The adjuvant chemotherapy is a minimally invasive technique. It consists of the administration of Idarubicin (Zavedos®, Pfizer) mixed with Lipiodol (Lipiodol Ultra-Fluid®, Guerbet) in the hepatic artery.The first course of treatment will be performed under general anesthesia at the same time as the percutaneous tumour ablation. The second and third cures will be performed under local anesthesia 3 and 6 weeks after percutaneous tumour ablation respectively. In the case of incomplete treatment during the percutaneous tumour ablation, the second intervention will be scheduled at the same time as the second intra-arterial chemotherapy treatment, under general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Age above 18 and under 80 years-old
* Chronic or histologically proven stage F3 or F4 hepatopathy, with liver hardness ≥ 10 kPa, or with imaging morphology suggestive of cirrhosis or portal hypertension
* Child-Pugh score ≤ B7
* Patients whose biological parameters meet the following criteria:

  * Platelets > 50,000 / mm3
  * Neutrophils > 1000 / mm3
  * Prothrombin ratio > 50%
  * Creatinemia < 150 μmol / L
  * Total bilirubinemia < 5 mg / dL
  * α-fetoprotein < 200 ng / mL
* Performance level of 0 or 1 according to "World Health Organization Performance Status"
* Presence of a single hepatocellular carcinoma of less than 3 cm with typical imaging characteristics as recommended by the American Association for the Study of Liver Diseases (AASLD)
* Patient with an indication of percutaneous tumor ablation (radiofrequency or microwave) under ultrasound or tomodensitometric identification
* Absence of heart failure (Left Ventricular Ejection Fraction (LVEF) > 50%)
* Women of childbearing age, using an effective method of contraception for the duration of treatment and at least 3 months after stopping the treatment.
* Male using an effective method of contraception throughout the treatment and at least 3 months after stopping the treatment

Exclusion Criteria:

* Presence on the initial imaging assessment of a macroscopic vascular invasion (portal or hepatic vein)
* Presence on initial imaging assessment of extrahepatic localization of hepatocellular carcinoma
* Presence of another untreated cancer
* Patients who previsouly received sphincterotomy or bilio-digestive anastomosis
* Contraindication to performing a general anesthesia
* Contraindication to performing an MRI scan
* Allergy to anthracyclines, iodine or gadolinium
* Contraindication to the injection of gadolinium-based contrast media.
* Contraindication to iodinated contrast agents
* Contraindication to Idarubicin (hypersensitivity to the active substance or excipients, severe heart disease, severe arrhythmia, severe renal or hepatic impairment, yellow fever vaccine or any other live attenuated vaccine for 6 months after discontinuation of chemotherapy, persistent myelosupressure, previous treatments with idarubicin and / or other anthracyclines or anthracenediones at maximum cumulative doses, mucositis, breastfeeding, uncontrolled infections, severe heart failure, myocardial infarction less than 6 months old).
* Contraindication to Lipiodol (Hypersensitivity, Hyperthyroidism, traumatic lesions, haemorrhage or recent bleeding)
* Patients who have already received or exceeded the recommended cumulative dose for anthracyclines (Idarubicin = 150 mg / m²)
* Patients who cannot temporarily stop their anticoagulant treatment or anti-platelet agent for the duration of the procedure
* Failure of endoscopic eradication of oesophageal varices of grade > 1
* Inability to adhere to the protocol
* Simultaneous participation to another clinical trial
* Patients not covered by health insurance

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2021-07-14 (Actual); Study Completion 2021-07-14 (Actual)

PRIMARY OUTCOMES:
The survival rate without hepatic recurrence at 1 year | 1 year
  Hepatic recurrence will be defined as the appearance on at least one hepatic MRI with gadolinium injection of a large diameter tumor site at least greater than 10 mm, and presenting characteristics of CHC (hyper vascularization at arterial time and washing at portal or late time), either at the edge of the percutaneous tumor destruction site (= local recurrence) or at a distance from the percutaneous tumor destruction site (= intrahepatic recurrence distant), or both, after at least one liver MRI scan with gadolinium injection showed the absence of tumor residues. Lesions of more than 10 mm that do not present with the typical CHC enhancement described above will be considered CHCs if they have a growth in size of at least 1 cm on successive controls.

SECONDARY OUTCOMES:
The incidence rate of local tumor recurrence | 1 to 2 years
  The incidence rate of local tumor recurrence at 1 and 2 years, defined as the appearance, on at least one hepatic MRI with gadolinium injection, of a tumor site with hepatocellular carcinoma characteristics at the edge of the percutaneous tumor ablation site.
The incidence rate of intrahepatic recurrence | 1 to 2 years
  The incidence rate of intrahepatic recurrence at 1 and 2 years defined as the appearance, on at least one hepatic MRI with gadolinium injection, of a tumor site with hepatocellular carcinoma characteristics at a distance from the percutaneous tumor ablation site.
The incidence rate of hepatic recurrence | 2 years
  The incidence rate of hepatic recurrence at 2 years defined as the appearance, on at least one hepatic MRI with gadolinium injection, of a tumor site with hepatocellular carcinoma, after at least one exploration by hepatic MRI with gadolinium injection, showed the absence of tumor residue.
Survival without hepatic recurrence | 2 years
  Survival without hepatic recurrence defined as the time between the date of randomization and the date of liver MRI, having confirmed, after centralized and blind re-examination, the presence of a hepatic tumor recurrence either local or intra distant hepatic. Patients who are deceased or transplanted will be considered to have liver progression at the time of death or transplantation.
Rate of survival without hepatic recurrence | 1 to 2 years
  Rate of survival without hepatic recurrence at 1 and 2 years defined as the absence of appearance of a large diameter tumor site (at least greater than 10 mm), presenting characteristics of hepatocellular carcinoma on the border of the percutaneous tumour ablation site.
Overall survival | 2 years
  Overall survival defined as the time between the date of randomization and the date of death of the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Christophe CASSINOTTO, Principal Investigator — University Hospital, Montpellier
Locations (1):
- UH Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No